CLINICAL TRIAL: NCT03158571
Title: Chilean Gastric Cancer Task Force (FORCE 1): A Study Protocol to Obtain a Clinical and Molecular Classification of a Cohort of Gastric Cancer Patients.
Brief Title: Chilean Gastric Cancer Task Force (FORCE 1)
Acronym: FORCE-1
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Center of Excellence of Precision Medicine (CEMP) (Unknown); Advanced Center for Chronic Diseases (ACCDiS) (Unknown); Millennium Institute on Immunology and Immunotherapy (Other); Center UC for Investigation in Oncology (CITO) (Unknown); Centre of Clinical Research, Health Technology Assessment Unit (Unknown); National Scientific and Technical Research Council (CONICET), Argentina (Unknown); Grupo Oncologico Cooperativo del Sur (GOCS), Argentina (Unknown); Hospital Universitario central de Asurias, Oviedo, España (Unknown); Hospital Morales Meseger, Murcia, España (Unknown); Centro de Cancer. Pontificia Universidad Católica de Chile (Unknown); Hematology and Oncology Department (Unknown)
Responsible Party: Sponsor
Other Study IDs: GCTF1
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Biomarkers
Keywords: Gastric Cancer; gastric adenocarcinoma; cancer subtypes; prognosis; survival; molecular classification; chemotherapy; immunotherapy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — RNA and DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background. Gastric cancer (GC) is the world's second leading cause of neoplastic mortality. Genetic alterations, response to treatments and mortality rates are highly heterogeneous across different regions. In Chile, GC is the leading cause of cancer death, affecting 20 per 100,000 people and >3,000 deaths/year. Clinical outcomes and response to "one size fits all" therapies are highly heterogeneous and thus a better stratification of patients may aid cancer treatment and response.

Study design/methods. The Gastric Cancer Task Force (GCTF) is a Chilean collaborative, non-interventional retrospective study that seeks to stratify gastric adenocarcinomas (GACs) using retrospect clinical outcomes and genomic, epigenomic and protein alterations in a cohort of 200 patients. Tumor samples from the pathology department and the Cancer Center at UC Christus healthcare network at Pontificia Universidad Católica de Chile will be analyzed using a panel of 143 known cancer genes (Oncomine Comprehensive Assay) at the Center of Excellence of Precision Medicine (CEMP) in Santiago, Chile. Additionally, gene promoter methylation will be performed and selected clinically relevant proteins (e.g. PD-L1, Erb-2, VEGFR2 among others) will be assessed by Tissue Microarray, Epstein-Barr virus (EBV) status will also be assessed. Observations will be correlated to 120 clinical parameters, including general patient information, cancer history, laboratory studies, comorbidity index, chemotherapy, targeted therapies, efficacy and follow-up.

Discussion. The development of a clinically meaningful classification that encompasses comprehensive clinical and molecular parameters may improve patient treatment, predict clinical outcomes, aid patient selection for clinical trials and offer insights into future preventive and/or therapeutic strategies.

DETAILED DESCRIPTION:
Participating entities: The Chilean Gastric Cancer Task Force (GCTF) is a collective effort between two principal identities: 1- The Center of Excellence of Precision Medicine (CEMP), which was established through a joint funding by the government agency for economic development (Corporacion de Fomento de la Produccion, CORFO) and Pfizer Chile and 2- The Center UC for Investigation in Oncology (CITO) based at the Pontificia Universidad Católica de Chile. Both entities are non-profit research organizations aimed at enhancing public education and implementing strategies to improve clinical outcomes in oncology treatment and cancer prevention.

Primary objective: To stratify Chilean GC patients into prognostic subgroups, and to correlate therapy response according to clinical, protein, epigenetic and genetic alterations in a cohort of 200 GAC patients.

Secondary objectives

* To determine the mutation profile in Chilean GC patients.
* To assess the percentage of Chilean GC patients that could benefit from currently available druggable targets (actionable genes).
* To correlate EBV presence to clinical parameters.
* To assess the expression levels of proteins associated with molecular stratifications and currently targeted therapies (eg. PD-L1 and antiangiogenics)
* To determine the profile of SNPs in the DPYD and TYMS genes in Chilean GC patients and their correlation with adverse events.

Study design

Ethics approval The GCTF is a non-interventional, collaborative, prospective non-concurrent study that seeks to stratify GAC patients based on their prognosis and therapy response. The study will strictly adhere to all legal requirements, regulations and general principles established by international agencies governing the ethical conduct in biomedical research on human subjects, following the good clinical practices and the declaration of Helsinki. The GCTF study protocol has been approved by the Ethics Committee of the University hospital (Pontificia Universidad Catolica de Chile , CEC MED UC approval number 16-046, resolution dated April 21st, 2016).

Patient recruitment & characteristics Diagnosed GC patients will be recruited from the Red UC Christus network in Santiago, Chile. Patient recruitment and signing of informed consent forms, maintenance and monitoring of patient medical records, biological material and sample extractions will be managed by CITO.

Patient and treatment history reveals that besides surgery and chemotherapy, approximately 10% of patients received Trastuzumab (ERBB2 targeted therapy, also called Herceptin), another 10% received immunotherapy including pembrolizumab and Ipilimumab (checkpoint inhibitors). Finally approximately 5% of patients received antiangiogenic therapy (consisting of VEGFR2 targeted therapy with Ramucirumab). Additionally, histological analysis showed that approximately 50% of patients were classified as intestinal type, 30% as diffuse, and 20% were either mixed or undetermined.

Inclusion criteria

* Adult male or female, aged >18 years
* Diagnosed with gastric cancer (histological or cytological)
* Attending health centers of the Red UC Christus network for at least 3 months with clinical follow-up
* Capable to read and speak Spanish
* Willing and able to provide written informed consent to the study that should be dated and signed at the time of enrollment.

Exclusion criteria

Patients:

* With small biopsy samples insufficient for analysis.
* Whose medical records cannot be collected or are unavailable.
* Without signed informed consent.

Clinical data Clinical data from patients will be obtained by healthcare providers and entered into an online electronic platform. Samples will be coded and patient identity known only to the attending physician. Clinical variables are divided into sections: General Patient Information, Cancer History, Laboratory Studies, Comorbidity (Charlson) Index, Chemotherapy, Efficacy & Follow Up and Toxicity. Patient chemotherapy will be classified by: regime, number of cycles & time of treatment and chemotherapy dose-intensity during the first 6 months. Chemotherapy regimens representing the first line chemotherapy prescribed to the patients. Full chemotherapy dose intensity during the first 6 months will be obtained through patient interviews and entered directly into the online platform. Finally, efficacy & follow-up and toxicity data obtained from patients.

Main clinical outcomes Main outcomes will be inferred from obtained clinical data, these include overall survival, progression-free, and recurrence-free survival rates.

Biological samples & Oncomine Comprehensive Assay Biological materials obtained at the Red UC Christus will be transported to CEMP in Santiago de Chile under standardized protocols. A total of 200 patient tumor samples will be obtained from archived Formalin Fixed Paraffin Embedded (FFPE) samples. Nucleic acids will be extracted using the RecoverAll kit (Thermo Fisher Cat #AM1975) and analyzed using the commercially available Oncomine Comprehensive Assay kit. This assay simultaneously analyzes DNA and RNA from samples allowing the assessment of 73 gene hotspots (based on DNA), 49 focal copy number variations (CNVs, DNA based), 26 full coding sequences (for mutations and CNV loss), and 22 gene fusion drivers (RNA). Notably, 72 of these genes are drug targets. Genomic raw data obtained (.vcf and .pdf files) will be stored and backed up in a local Data Center for subsequent genomic analysis. Upon publication of the findings of this study, the Oncomine results along with clinical classification of individual tumors will be made publicly available.

Tissue Micro Array (TMA) Analysis The following genes will be further analyzed by a TMA using specific antibodies against: PD-L1 (Dako, Cat # SK00521), PD-L2 (Thermo Cat# B7-DC/CD273), Phosphorylated mTOR (Abcam Cat#AB118815), p53 (Cat # 5278074001), VEGFR2 (Abcam Cat #AB39256), Phosphorylated Akt (Thermo Cat #473), HER2 (Roche, Cat # 05278368001), p16 (Roche, Cat # 06695221001), Met (Abcam Cat #AB51067), HA-4 (Abcam Cat #AB24480) and four microsatellite markers (all from Roche): MLH1 (Cat # 06472966001), MSH2 (Cat # 05269270001), MSH6 (Cat # 5929911001), PMS2 (Cat # 06419216001). Manual TMA will be prepared as described previously. Briefly, paraffin blocks will be obtained and cut and stained by Hematoxylin & Eosin (H&E) in order to select the best histological area. Subsequently selected tissue area will be placed into the TMA by circling the identified area in the corresponding block. Cylindrical core biopsies will be extracted from each paraffin block using a 1 mm stylet and placed into a new recipient block. Selected adequate cases had tumors that occupied at least 10% of the core area. Each case will be processed in triplicate to prevent tissue loss during cutting. Sections from each tissue array block will be cut, de-paraffinized and dehydrated for H&E and immunohistochemical procedures.

Gene methylation Promoter gene methylation on six selected genes that have previously shown promoter regulation by methylation associated with GC will be assessed. Methylation analysis will include the reprimo gene and other mRNAs associated with GC progression. Analysis will be performed by bisulfite sequencing as described previously using the EZ DNA methylation Gold kit (Zymo Research) with minor modifications. Briefly, bisulfite treated DNA is amplified using specific PCR primers, with PCR products subsequently cloned and sequenced.

EBV identification EBV subtypes in patient samples will be assessed using the chromogenic in situ hybridization (CISH) method with minor modifications.

Single Nucleotide Polymorphism (SNP) analysis A significant proportion of GC patients can develop serious toxicity from 5-FU treatment including bone marrow suppression, neuropathy, low white blood cell numbers, fever, infections, nausea, vomiting, severe diarrhea, mouth and digestive tract inflammation, all of which are recorded in the patient history of other cohorts. Subtle personal and population changes in DNA, called SNPs can account for increases in the risk of 5-FU toxicity; 5-FU metabolism is predominantly hepatic, where the enzyme DPYD is responsible for metabolizing >80% of the drug, producing the inactive metabolite 5,6 dihydroxy-5-FU. It is widely documented that a decreased DPYP activity is associated with severe toxicity. Non-metabolised fraction of 5-FU (20%) is transformed by a series of enzymes (e.g TP, TK), producing the active metabolites that will cause TYMS inhibition, thereby promoting DNA/RNA damage. Variations in TYMS and MTHFR genes (related to reduced folate synthesis, increased 5-FU effect), have been associated with toxicity by treatment with 5-FU. The approach that was used to select the genetic variants consisted of a search in the database, PharmGKB. A total of six non-synonymous SNPs will be analyzed: four of them comprise the DPYD gene, one for TYMS and one for MTHFR. Analysis will be performed using TaqMan™ SNP Genotyping Assay technology (Applied Biosystems™). SNPs will be assessed in DNA isolated from paraffin embedded patient samples.

Sample size and statistical analysis

The minimum sample number will be calculated in order to ensure the goals of the project are fully accomplished. Considering that approximately 90% of GC cases are indeed GAC, at 5% error rate and at 95% confidence interval the investigators originally projected a sample size of 200 patients. However the investigators have also considered a 15% rate of sample loss (defective samples or patient drop-out), which gave a total of 230 patients to be recruited.

Standard descriptive statistics will be utilized to analyze qualitative and quantitative variables, such as relative and absolute frequencies, frequency tables, average, median, standard deviation, range and quartiles. A 95% confidence will be considered appropriate for analysis. Descriptive statistics will also be used to characterize the most relevant clinical parameters measured. The association of categorized variables will be performed by chi-square or Fisher's exact tests. One arm Analysis of Variance will compare continuous variables among groups. Survival outcome studies will be accomplished using the Kaplan-Meier method. Prognostic factors will be evaluated according to the Cox proportional hazards regression model.

Principal component analysis (PCA) of the genes variants will be conducted and the association of the first principal components with a small pre-defined set of genomic alteration signatures will be assessed. To define molecular subgroups, the investigators will utilize unsupervised clustering. The correlation of the molecular subtypes with clinical data (e.g. age, gender, Lauren class) and clinical outcomes (e.g. overall survival, response rate) will be assessed. Moreover, supervised classification will be performed based on clinical outcomes and the resulting groups of both approaches will be compared with other reported molecular subtypes.

Patient protection/written informed consent forms

All parties guarantee the protection of the patients' personal records. Patient names are not included in any form in sheet-reports, publications, or in any type of publishable document derived from the study with the exception of documents required by law. Informed consent forms are elaborated strictly following legal and local regulations. The written informed consent forms, including all changes made throughout the study must be prospectively approved by the Internal Review Board/independent Ethics Committee, and CEMP prior to be incorporated into the study.

The investigators, representatives or healthcare providers will obtain written informed consent forms from every patient or a legal representative before any specific activity of the study is performed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with gastric cancer (histological or cytological) Attending health centers of the Red UC Christus network for at least 3 months with clinical follow-up.

Capable to read and speak spanish Willing and able to provide written informed consent to eh study that should be dated and signed informed consent

Exclusion Criteria:

* With small biopsy samples insufficient for analysis. Whose medical records cannot be collected or are unavaible Without signed informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chilean population diagned with gastric cancer
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | two years
  Overall survival of patients with gastric cancer

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Garrido, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Yes
Public information of the data base
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available within 6 months after study completion.
Access Criteria: Access request will be reviewed by the principal investigator.

REFERENCES:
- [Derived] Cordova-Delgado M, Pinto MP, Retamal IN, Munoz-Medel M, Bravo ML, Fernandez MF, Cisternas B, Mondaca S, Sanchez C, Galindo H, Nervi B, Ibanez C, Acevedo F, Madrid J, Pena J, Koch E, Maturana MJ, Romero D, de la Jara N, Torres J, Espinoza M, Balmaceda C, Liao Y, Li Z, Freire M, Garate-Calderon V, Caceres J, Sepulveda-Hermosilla G, Lizana R, Ramos L, Artigas R, Norero E, Crovari F, Armisen R, Corvalan AH, Owen GI, Garrido M. High Proportion of Potential Candidates for Immunotherapy in a Chilean Cohort of Gastric Cancer Patients: Results of the FORCE1 Study. Cancers (Basel). 2019 Aug 30;11(9):1275. doi: 10.3390/cancers11091275. PMID 31480291
- [Derived] Owen GI, Pinto MP, Retamal IN, Fernadez MF, Cisternas B, Mondaca S, Sanchez C, Galindo H, Nervi B, Ibanez C, Acevedo F, Madrid J, Pena J, Bravo ML, Maturana MJ, Cordova-Delgado M, Romero D, de la Jara N, Torres J, Rodriguez-Fernandez M, Espinoza M, Balmaceda C, Freire M, Garate-Calderon V, Crovari F, Jimenez-Fonseca P, Carmona-Bayonas A, Zwenger A, Armisen R, Corvalan AH, Garrido M. Chilean Gastric Cancer Task Force: A study protocol to obtain a clinical and molecular classification of a cohort of gastric cancer patients. Medicine (Baltimore). 2018 Apr;97(16):e0419. doi: 10.1097/MD.0000000000010419. PMID 29668600